CLINICAL TRIAL: NCT06130254
Title: Phase Ib Trial of the KRAS G12C Inhibitor Adagrasib (MRTX849) in Combination With the PARP Inhibitor Olaparib in Patients With KRAS G12C Mutated Advanced Solid Tumors, With a Focus on Gynecological, Breast, Pancreatic and KEAP1 Mutated Non-small Cell Lung Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0136; NCI-2023-09685 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumor; Non-small Cell Lung Cancers
MeSH Terms: interventions — adagrasib; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adagrasib+Olaparib (Experimental): Participants will take adagrasib and olaparib by mouth 2 times each day. Each dose should be taken at about 12 hours apart (1 dose in the morning, 1 dose in the evening). The study drugs should be swallowed whole with water. Do not chew, crush, dissolve, or divide the study drugs.
  If forget a dose and less than 2 hours have passed since the usual time participants take the study drug, take the dose as soon as participants remember. If more than 2 hours have passed, do not take the dose. Wait and take the next dose as scheduled
  Interventions: Drug: Adagrasib; Drug: Olaparib

INTERVENTIONS:
Drug: Adagrasib — Given by PO BID
  Other Names: MRTX849
Drug: Olaparib — Given by PO BID
  Other Names: Lynparza™

SUMMARY:
Evaluate safety and tolerability, while establishing the recommended dose of the investigational drug combination of adagrasib and olaparib that can be given to participants with advanced solid tumor(s) with a KRAS G12C and/or KEAP1 mutation.

DETAILED DESCRIPTION:
Primary Objectives

* To evaluate the safety and tolerability of adagrasib in combination with olaparib in participants with KRAS G12C mutant advanced solid tumors.
* To establish the maximum tolerated dose and/or recommended phase 2 dose (MTD/RP2D) of the combination in participants with KRAS G12C mutant advanced solid tumors.

Secondary Objectives

* To assess the preliminary antitumor activity of the combination of adagrasib in combination with olaparib using objective response rate (ORR) = RECISTv1.1 complete response plus partial response (CR+PR).

Exploratory Objectives

* To assess predictive biomarkers of response and resistance to the combination of adagrasib with olaparib.
* To evaluate the pharmacodynamic profile of the combination of adagrasib and olaparib in participants with KRAS G12C mutant advanced solid tumors.
* To assess potential mechanisms of response and resistance by comparing serially collected circulating tumor DNA (ctDNA) samples and biopsies in responders and non-responders.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥ 18 years old and must fulfil all the following inclusion criteria to be eligible for enrollment into the study.

  1. Dose escalation cohort: Histologically confirmed diagnosis of a solid tumor malignancy with a KRAS G12C mutation. Participants are eligible based on detection of these mutations in tumor tissue or plasma circulating tumor DNA (ctDNA) with a minimum VAF of 1%.
  2. Dose expansion cohort 1: Histologically confirmed diagnosis advanced pancreatic cancer with KRAS G12C mutation. Participants must have progressed on at least 1 prior line of standard systemic therapy and must be eligible based on detection of KRAS G12C mutation in tumor tissue or ctDNA with a minimum VAF of 1%.
  3. Dose expansion cohort 2: Histologically confirmed diagnosis of advanced breast cancer with KRAS G12C mutation. Participants must have progressed on at least 1 prior line of standard systemic therapy and must be eligible based on detection of KRAS G12C mutation in tumor tissue or ctDNA with a minimum VAF of 1%.
  4. Dose expansion cohort 3: Histologically confirmed diagnosis of advanced uterine or epithelial ovarian cancer with KRAS G12C mutation. Participants must have progressed on at least 1 prior line of standard systemic therapy and must be eligible based on detection of KRAS G12C mutation in tumor tissue or ctDNA with a minimum VAF of 1%.
  5. Dose expansion cohort 4: Histologically confirmed diagnosis of NSCLC with KRAS G12C and KEAP1 co-mutations. Participants must have progressed on at least 1 prior line of standard systemic therapy and must be eligible based on detection of KRAS G12C and KEAP1 co-mutations in tumor tissue or plasma circulating tumor DNA (ctDNA) with a minimum VAF of 1%.
  6. Unresectable or metastatic disease and for which standard curative or palliative measures do not exist or are no longer effective.
  7. Participants must have evaluable or measurable disease per RECIST v1.1 for the dose escalation cohort and must have measurable disease per RECIST v1.1 for dose expansion cohorts 1-4.
  8. Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
  9. Life expectancy of at least 3 months.
  10. Most recent prior systemic therapy (e.g., chemotherapy, immunotherapy or, investigational agent) and radiation therapy discontinued at least 2 weeks before first dose date.
  11. Eastern Cooperative Oncology Group (ECOG) performance status in 0 or 1 (see Appendix 1).
  12. Laboratory values within the screening period:

      1. Absolute neutrophil count ≥ 1.5 x 109/L
      2. Platelet count ≥ 100,000/mm3 (≥ 100 x 109/L)
      3. Hemoglobin ≥ 10 g/dL, in the absence of transfusions for at least 28 days
      4. Total bilirubin ≤ 1.5 x Upper Limit of Normal (ULN) (if associated with liver metastases or Gilbert's disease, ≤ 3 x ULN)
      5. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN (if associated with liver metastases, ≤ 5 x ULN)
      6. Creatinine clearance ≥51mL/min calculated using a validated prediction equation:

      Estimated GFR= (140-age(years)∙ Weight (Kg)∙F)/(serum creatine (mgdL)∙72), where F=0.85 for females and F=1 for males.
  13. The effects of adagrasib on the developing human fetus are unknown. For this reason and because the therapeutic agents used in this trial are known to be teratogenic, women and men, who are sexually active and of childbearing potential, must agree to use two highly effective forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 6 months following termination of the study treatment (MDA Policy CLN 1114). This includes all female participants, between the onset of menses between 18 and 55 years, unless the patient presents with an applicable exclusionary factor which may be one of the following: (i) Postmenopausal (no menses in greater than or equal to 12 consecutive months); (ii) History of hysterectomy or bilateral salpingo-oophorectomy; (iii) Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy); (iv) History of bilateral tubal ligation or another surgical sterilization procedure; (v) radiation-induced oophorectomy with last menses at least 1 year ago; and (vi) chemotherapy-induced menopause with at least 1 year interval since last menses. Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
  14. Men treated or enrolled on this protocol must also agree to use adequate contraception and avoid donating sperm prior to the study, for the duration of study participation, and 6 months after completion of the trial.
  15. Prior treatment with a therapy targeting PARP or KRAS G12C mutation is permitted.
  16. Ability to understand and the willingness to sign a written informed consent document.
  17. Willing to comply with clinical trial instructions and requirements.

Exclusion Criteria:

* Participants presenting with any of the following will not be included in the study:

  1. Active brain metastases. Patients are eligible if brain metastases are adequately treated and patients are neurologically stable (which is assessed in a case-by-case by the treating physician based on the likelihood of central nervous system (CNS) activity - except for residual signs or symptoms related to the CNS treatment- and by the lack of corticosteroid dosing or by having a stable or decreasing dose of ≤ 10 mg daily prednisone, or equivalent) for at least 2 weeks prior to enrollment.
  2. Participants with carcinomatous meningitis.
  3. Participants with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of MDS/AML.
  4. Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1), excluding alopecia.
  5. History of significant hemoptysis or hemorrhage within 4 weeks of the first dose date.
  6. Undergone major surgery within 4 weeks of first dose date, or not recovered from any major surgery that occurred >2 weeks before starting study treatment.
  7. Undergone allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
  8. History of intestinal disease, inflammatory bowel disease, major gastric surgery, or other gastrointestinal conditions (e.g., uncontrolled nausea, vomiting, malabsorption syndrome) likely to alter absorption of study treatment or result in inability to swallow oral medications.
  9. Any of the following cardiac abnormalities:

     1. Unstable angina pectoris or myocardial infarction within 6 months prior to enrollment
     2. Congestive heart failure NYHA ≥ Class 3 within 6 months prior to enrollment
     3. Left ventricular ejection fraction (LVEF) < 50%
     4. QTc > 480 milliseconds or medical or immediate family history of congenital Long QT Syndrome
     5. Symptomatic or uncontrolled atrial fibrillation or other arrhythmia within 6 prior to enrollment
     6. History of uncontrolled ventricular arrhythmia, recent (within 6 months) myocardial infarction
  10. History of stroke or transient ischemic attack within 6 months prior to enrollment.
  11. Concomitant use of known strong CYP3A inhibitors or moderate CYP3A inhibitors listed in Section 5.5 and Appendix 4, Table 23. The required washout period prior to starting study treatment is 2 weeks.
  12. Concomitant use of known strong or moderate CYP3A inducers listed in Section 5.5 and Appendix 4, Table 23. The required washout period prior to starting study treatment is 5 weeks.
  13. Use of a medication with any of the following characteristics, which cannot be switched to an alternative treatment prior to study entry:

      1. Substrate of P-gp with narrow therapeutic index
      2. Strong inhibitor of BCRP
      3. Proton pump inhibitor
      4. Known risk of QT prolongation or Torsades de Pointes
      5. Any substances listed in Section 6.3
  14. Known or suspected presence of another malignancy, unless curatively treated, with no evidence of disease for ≥5 years with the exception of adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1-grade 1 endometrial carcinoma.
  15. Known history of human immunodeficiency virus (HIV) infection or acute or chronic

      Hepatitis B or C infection. Note that the following are permitted:
      1. Participants treated for hepatitis C with no detectable viral load;
      2. Patients treated for HIV with no detectable viral load for at least 1 month prior to enrollment while on a stable regimen of agents that are not strong inhibitors of CYP3A4
  16. Pregnancy. WOCBP must have a negative serum or urine pregnancy test documented within the 28-day screening period prior start of study drug.
  17. Breast-feeding or planning to breast feed during the study or within 6 months after study treatment.
  18. Any serious illness, uncontrolled inter-current illness, psychiatric illness, active or uncontrolled infection, or other medical history, including laboratory results, which, in the Investigator's opinion, would be likely to interfere with the participant's participation in the study, or with the interpretation of the results.
  19. History of uncontrolled ventricular arrhythmia, recent (within 6 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan
  20. Participants with a known hypersensitivity to olaparib or any of the excipients of the product
  21. Patients that received live virus and live bacterial vaccines within 3 days of trial enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2028-08-25 (Estimated); Study Completion 2030-08-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Yap, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org